CLINICAL TRIAL: NCT04109807
Title: Effects of Low Dose Ozone on Airway Inflammatory Responses in Adults With Asthma Asthma SNOZ
Brief Title: Effects of Low Dose Ozone on Airway Inflammatory Responses in Adults With Asthma - Sedentary Nasal Ozone (Asthma SNOZ)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment for this study was stopped due to Covid and will resume once it is determined acceptable to do inhalational challenges. rebuilding chambers after EPA was shut down.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); North Carolina State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-2425
Record Dates: First submitted 2019-09-23; First posted 2019-09-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Asthma, Allergic
MeSH Terms: conditions — Asthma | interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6 hour Filtered Air (FA) followed by O3 exposure (Experimental): For the first exposure session, participants are exposed to filtered air (FA) for 6 hours. For the second exposure session, the same participant will be exposed to ozone at a concentration of 0.07ppm for 6 hours.
  Interventions: Other: Ozone; Other: FA
- 6 hour O3 exposure followed by FA exposure (Experimental): For the first exposure session, a participant will be exposed to ozone at a concentration of 0.07ppm for 6 hours. For the second exposure session, the same participant will be exposed to FA for 6 hours.
  Interventions: Other: Ozone; Other: FA

INTERVENTIONS:
Other: Ozone — ozone exposure
Other: FA — Filtered air exposure

SUMMARY:
To determine if low levels of ozone (O3) encountered on a typical day in Chapel Hill will decrease spirometric values in mild asthmatics.

DETAILED DESCRIPTION:
Short-term exposure to ambient air ozone has been recognized for decades to be adversely associated with impacts on the respiratory system. Indeed the evidence is such that the Environmental Protection Agency (EPA) has determined that there is a causal relationship, and even lowered the 8-hour exposure standard to 0.07 parts per million (ppm) in 2015. Controlled human exposure studies and epidemiological studies have consistently observed ozone-associated decrements in lung function and increased respiratory symptoms. Most controlled human exposure studies have been performed with high ozone concentrations. Additionally, epidemiologic studies have focused on populations engaged in outdoor activities (increasing ozone exposure through increased minute ventilation), or in cities such as Los Angeles or Mexico City where ambient ozone levels are especially high. Evidence has recently emerged that exposure to low ozone concentrations also produces adverse health effects, especially among susceptible groups including children with asthma.

The objective of this study is to examine if low level ozone exposure (compared to a clean air exposure), reflective of a typical metropolitan summer day, will cause decrements in lung function and measurable upper and lower airway inflammation in mild asthmatics (who are not on asthma controller medications) while performing typical daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45, both sexes included
* Mild intermittent asthma, defined as daytime asthma symptoms no more than 2 times per week, night time asthma symptoms no more than 2 times per month, FEV1 >80% of predicted, and asthma exacerbation requiring oral steroids 1 time or less per year.
* Good general health as evidenced by medical history
* Vital signs will be within normal limits on admission to the study: oxygen saturation by pulse oximetry (SpO2) > 94%, systolic blood pressure between 150-90 mm Hg, diastolic blood pressure between 100-60 mm Hg, afebrile.
* FEV1 of at least 80% of predicted at baseline
* Able to provide informed consent
* Proof of Covid Vaccination

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes, chronic renal disease, chronic thyroid disease, history of chronic infections/immunodeficiency, history of tuberculosis
* Physician directed emergency treatment for an asthma exacerbation within the preceding 12 months
* Orthopedic injuries or impediments that would preclude bicycle or treadmill exercise
* Viral upper respiratory tract infection within 4 weeks of challenge.
* Any acute infection requiring antibiotics within 4 weeks of exposure or fever of unknown origin within 2 weeks of challenge.
* Individuals who use daily controller medication for asthma. Pre-treatment with a short acting bronchodilator prior to exercise is allowed.
* Nasal surgery within 6 months
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* Any recent or current use of nicotine
* History of intubation for asthma
* Pregnancy or nursing an infant as EPA strictly prohibits intentional exposure for research to this population.
* Covid infection in the past 90 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Percent (%) predicted forced expiratory volume at one second (FEV1) | 6 hours post-O3 versus post-air exposure versus pre-exposure
  Change from baseline %predicted FEV1 post-O3 versus post-air exposure.

SECONDARY OUTCOMES:
Change in Percent (%) predicted forced vital capacity (FVC) | 6 hours post-O3 versus post-air exposure versus pre-exposure
  Change from baseline %predicted FVC post-O3 versus post-air exposure.
Change in Percent eosinophils in induced sputum | 24 hours post-O3 versus post-air exposure
  % eosinophils in induced sputum (24 hrs post ozone - post air)
Change in Percent (%) neutrophils in induced sputum | 24 hours post-O3 versus post-air exposure
  % neutrophils in induced sputum (24 hrs post ozone - post air)
Change in Eosinophils per mg of induced sputum | 24 hours post-O3 versus post-air exposure
  Eosinophils per mg of induced sputum (24 hrs post ozone - post air)
Change in neutrophils per mg of induced sputum | 24 hours post-O3 versus post-air exposure
  Neutrophils per mg of induced sputum (24 hrs post ozone - post air)
Change in Cytokine concentrations in induced sputum picograms per milliliter (pg/mL) | 24 hours post-O3 versus post-air exposure
  Cytokine and via Mesoscale in induced sputum (pg/mL)
Change in Cytokine concentrations in Nasal Epithelial Lining Fluid (NELF) | 6 hours post-O3 versus post-air exposure
  Cytokine via Mesoscale in NELF
Change in Change in cytokine concentrations in Nasal Epithelial Lining Fluid (NELF) | 24 hours post-O3 versus post-air exposure
  Cytokine and via Mesoscale in NELF
Change in Fraction of Exhaled Nitric Oxide (FENO) levels in parts per billion (PPB) | 6 post-O3 post-air exposure versus pre-exposure
  Changes in FeNO levels in ppb (6 hours post ozone - post air)
Change in FENO levels in parts per billion (PPB) | 24 hours post-O3 versus post-air exposure
  Changes in FeNO levels in ppb (24 hours post ozone - post air)

CONTACTS AND LOCATIONS:
Overall Officials: David Peden, MD, Principal Investigator — UNC SOM
Locations (1):
- University of North Carolina CEMALB, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: Approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.